CLINICAL TRIAL: NCT04426227
Title: The Effect of Gaze Training on Task Performance and Skill Acquisition in Ultrasound-guided Regional Anaesthesia: a Partially Blinded Randomised Controlled Trial.
Brief Title: Gaze Training on Task Performance Regional Anaesthesia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, David Hewson, Honorary Assistant Professor, University of Nottingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 434-1912
Record Dates: First submitted 2020-06-02; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Anesthesia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Gaze (Experimental): The gaze-trained group will be shown a video, derived from the eye tracker, of an expert's visual control whilst performing the ultrasound task. Participants will be made aware of the target-focused gaze strategy (lengthy and stable fixations on the needling target), and the manner in which the gaze shifted from target to tools (hands, needle and transducer) in a fast, smooth fashion. They will then be advised to try to mimic the gaze strategy of the expert while undertaking the needling task as their first training task. After completion of this training task, participants will be shown their own video data, as captured by the eye tracker. Participants will be asked to comment on differences between their own video and the expert video they had previously seen. This feedback process will be replicated a further four training task attempts. Participants in this group will therefore undergo a total of five training attempts of the needling task.
  Interventions: Other: Gaze training
- Group Discovery (Active Comparator): The discovery learning group will be given no video feedback and will be instructed to perform five training attempts at the needling task without further training or feedback.
  Interventions: Other: Discovery learning

INTERVENTIONS:
Other: Gaze training — A training module in gaze training for peripheral nerve blockade
  Arms: Group Gaze
Other: Discovery learning — A phase of discovery learning guided by novice operators themselves
  Arms: Group Discovery

SUMMARY:
Regional anaesthesia is the performance of spinal, epidural or peripheral nerve blocks to allow patients to undergo surgery awake and to provide post-operative pain relief. Anaesthetists inject local anaesthetic using specialist needles close to nerves to prevent transmission of pain. Hand-held ultrasound is often used by anaesthetists to direct these needles to the correct position i.e. close to, but not in the nerve itself. If the needle is not adequately seen using the hand-held ultrasound it may pierce the nerve causing permanent nerve damage and significant patient harm.

Within the time and resource constraints of postgraduate medical training, it would be advantageous to optimise expertise acquisition of practical skills with a cheap, self-directed educational intervention. Therefore, the aim of this study is to determine whether gaze training is associated with improved performance of an ultrasound-guided needle task. The investigators hypothesise that improved gaze control will translate to better technical performance of an ultrasound-guided regional anaesthesia task.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate Science, Technology, Engineering or Maths (STEM) students who are capable of giving informed consent

Exclusion Criteria:

* Previous experience of gaze training or eye tracking software
* Previous experience of regional anaesthesia needling tasks

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Composite Error Score | Undertaken during ultrasound assessment 1 (before training intervention) and during ultrasound assessment 2 (which will occur 10 minutes after the training intervention was undertaken). Each assessment will be 15 minutes in duration.
  Objective error scoring of performance at needling task

SECONDARY OUTCOMES:
Change in Global Rating Scale | Undertaken during ultrasound assessment 1 (before training intervention) and during ultrasound assessment 2 (which will occur 10 minutes after the training intervention). Each assessment will be 15 minutes in duration.
  Objective performance scoring of needling task, scored from 0-35, higher scores indicating better task performance.

OTHER OUTCOMES:
Change in Task completion time | Undertaken during ultrasound assessment 1 (before training intervention) and during ultrasound assessment 2 (which will occur 10 minutes after the training intervention was undertaken). Each assessment will be 15 minutes in duration.
  Time taken to finish needling task
Change in Fixation durations | Undertaken during ultrasound assessment 1 (before training intervention) and during ultrasound assessment 2 (which will occur 10 minutes after the training intervention was undertaken). Each assessment will be 15 minutes in duration.
  The total duration in seconds during the task that the participant spends engaging fixation visual behaviour in pre-defined areas of interest during the needling task

CONTACTS AND LOCATIONS:
Overall Officials: David W Hewson, MBBS, Principal Investigator — University of Nottingham

IPD SHARING:
Plan to Share IPD: No